CLINICAL TRIAL: NCT00871793
Title: Effect of Occupational Therapy on the Function and Mobility in Supracondylar Humerus Fractures: A Randomized Controlled Trial
Brief Title: Effect of Occupational Therapy on the Function and Mobility of Elbow Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Schmale, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AEF-24801
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Supracondylar Humerus Fracture
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Occupational therapy
  Interventions: Other: Occupational therapy
- 2 (No Intervention): watchful waiting

INTERVENTIONS:
Other: Occupational therapy — Participants in this arm will receive six sessions of occupational therapy in a 5 week period.
  Arms: 1

SUMMARY:
Supracondylar humerus fracture are common upper extremity injuries in children accounting for over 400 fractures per year and approximately 25% of all fractures treated at Seattle Children's Emergency Department. Most of these fractures are treated with splints and casts though more than one-third undergo surgical fixation followed by casting. Healing is usually complete after 3-4 weeks, when casts (and pins, if fixed operatively) are removed and motion begun. Though stiffness is often a problem after immobilization of adult elbow fractures, stiffness after pediatric elbow fractures is regarded as typically transient. This study addresses the question "Does early motion of the arm with physiotherapy promote the return of function and motion in patients with supracondylar humerus fractures?" The investigators will conduct a prospective randomized trial to determine the effect of six occupational therapy visits over a five week period of time on elbow function and mobility after supracondylar humerus fracture. The investigators will measure motion of the elbow and administer the child and parental Activity Scale for Kids performance versions (ASKp) assessment tool to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* Have a supracondylar fracture which is isolated, non - comminuted, and less than one week old.
* Will be treated with either casting or surgery.
* Lack head injuries or other fractures.
* Are not cognitively impaired or critically ill.
* Are 5 - 12 years old
* Speak English or Spanish

Exclusion Criteria:

* Requires open reduction to align
* Comminuted or t - intercondylar fracture
* Other fractures on the same limb
* Head injury
* Cognitive impairment
* Critically ill
* Mental disorders
* Fracture occurred more than one week prior to visit.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Activity Scale for Kids performance version (ASKp) | week 1, week 6, week 12, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Schmale, MD, Principal Investigator — University of Washington - Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States